CLINICAL TRIAL: NCT02918084
Title: A Phase III Study Comparing the Concurrent Versus the Sequential Administration of Chemotherapy and Aromatase Inhibitors, as Adjuvant Treatment of Post-menopausal Patients With Endocrine-responsive Early Breast Cancer.
Brief Title: CONcurrent vs SEqueNTial Adjuvant Treatments in Early Breast Cancer
Acronym: GIM10-CONSENT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Collaborators: Clinical Research Technology S.r.l. (Industry)
Responsible Party: Principal Investigator, Lucia Del Mastro,MD, Director of S.S. Innovative Therapies Unit, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIM10-CONSENT; 2013-001629-23 (EudraCT Number)
Record Dates: First submitted 2016-09-16; First posted 2016-09-28 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: sequential administration chemiotherapy; early breast cancer; breast cancer; aromatase inhibitor; adjuvant; post menopausal
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Letrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM A (Sham Comparator): Adjuvant chemotherapy → Aromatase inhibitors x 5 yrs (sequential arm)
  Interventions: Drug: Anastrozole or Letrozole or Exemestane
- ARM B (Experimental): Adjuvant chemotherapy + Aromatase inhibitors x 5 yrs (concurrent arm)
  Interventions: Drug: Anastrozole or Letrozole or Exemestane

INTERVENTIONS:
Drug: Anastrozole or Letrozole or Exemestane — Adjuvant chemotherapy → Anastrozole or Letrozole or Exemestane once a day for 5 years (sequential arm)
  Other Names: Clinical Practice
  Arms: ARM A
Drug: Anastrozole or Letrozole or Exemestane — Adjuvant chemotherapy + Anastrozole or Letrozole or Exemestane once a day for 5 years (concurrent arm)
  Other Names: Experimental arm
  Arms: ARM B

SUMMARY:
Breast cancer is the most common form of cancer among women. For patients candidated for adjuvant chemotherapy and endocrine therapy the optimal timing for their has not been clearly defined yet.

DETAILED DESCRIPTION:
Breast cancer is the most common form of cancer among women in North America, Europe and Latin America. Because nearly 80% of breast cancers are endocrine-responsive tumors, the majority of patients candidates for adjuvant chemotherapy (CT) are also candidates for endocrine therapy (ET). The optimal timing (i.e. concomitant vs sequential administration) for the integration of these two treatments has not been clearly defined yet.

In patients with hormone receptor positive early stage breast cancer who are candidates to adjuvant chemotherapy and endocrine therapy, the optimal timing for the integration of these two treatment modalities has not been clearly defined yet.

ELIGIBILITY:
Inclusion Criteria:

* Women with histological diagnosis of invasive breast cancer completely removed by surgery, any T, any N.
* Postmenopausal status defined by at least one of the following conditions:

  1. Aged ≥ 60
  2. Aged 45-59 and satisfying one or more of the following criteria:

     * amenorrhea for ≥12 months and intact uterus;
     * amenorrhea for <12 months and follicle-stimulating hormone (FSH) within the postmenopausal range, including:

       * pts with hysterectomy
       * pts who have received hormone replacement therapy (HRT)
       * pts with chemotherapy-induced amenorrhea
  3. bilateral oophorectomy at any age >18 years.
* Primary tumor positive for Estrogen Receptors (ER) and/or Progesteron receptors (PgR) (≥1% tumor cells positive by immunohistochemistry or ≥ 10 fmol/mg cytosol protein by ligand binding assay).
* Patients who are prescribed 5 years of endocrine therapy with an aromatase inhibitors (AI)
* Indication for adjuvant chemotherapy- Patients with HER-2 positive tumors are eligible provided that they are prescribed trastuzumab according to registered schedule.
* Signed informed consent.

Exclusion Criteria:

* HRT currently assumed or during the month before randomization
* Recurrent or metastatic disease
* HER-2 positive tumors if treatment with trastuzumab is considered not appropriate/feasible
* Concurrent illness that contraindicate adjuvant endocrine treatment and/or chemotherapy
* Patients who have received Tamoxifen as part of any breast cancer prevention trial
* Previous history of invasive breast cancer or other invasive malignancy within the previous 10 years, other than squamous or basal cell carcinoma of the skin or carcinoma in situ of the cervix, adequately cone biopsied
* Concomitant severe disease which would place the patient at unusual risk
* Concurrent treatment with experimental drugs
* Patients treated with systemic investigational drugs within the past 30 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2013-06; Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Disease- free Survival (DFS) | up to 15 years
  the primary outcome indicator will be the so called DFS, defined as time elapsing between the date of randomization and the date of one of the following events, whichever occurs first, assessed up to 15 years:
  * Local Recurrence of disease
  * Regional recurrence of disease
  * Distant recurrence of disease
  * Contralateral invasive or intraductal breast cancer
  * Second primary malignancy other than breast
  * Death for any cause

SECONDARY OUTCOMES:
Overall Survival (OS) | time between the date of randomization up to the date of death for any cause, assessed up to 15 years.
Translational Study: genomic analysis | up to 15 years
  Expression of genes associated with ER and Ki67 expression will be analyzed by Real Time polymerase chain reaction (PCR) on RNA extracted from formalin-fixed paraffin embedded (FFPE) sections of tumors classified as intermediate risk by clinical and pathological variables (stage I-II, G2, hormone receptors positive) and will be correlated with disease free survival.
Translational Study: epigenetic analysis | up to 15 years
  miRNA expression analysis by real time PCR and DNA methylation analysis by pyrosequencing will be assessed on FFPE sections of tumors classified as intermediate risk by clinical and pathological variables (stage I-II, G2, hormone receptors positive)
Translational Study: proteomic analysis | up to 15 years
  The different proteomic profiles identified in FFPE sections of hormone receptors positive G2 tumors will be correlated with DFS

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Del Mastro, MD, Principal Investigator — IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Locations (74):
- Italy (74):
  - Ospedale Santo SpiritoH, Casale Monferrato, AL
  - Ospedale di Rete 'Engles Profili' - A.S.U.R. Area Vasta 2, Fabriano, AN
  - A.O. San Giuseppe Moscati, Avellino, AV
  - Istituto Tumori 'Giovanni Paolo II' - IRCCS Ospedale Oncologico, Bari, BA
  - ASST Papa Giovanni XXIII - Ospedale Papa Giovanni XXIII, Bergamo, BG
  - Azienda Ospedaliera Treviglio-Caravaggio, Treviglio, BG
  - Azienda Ospedaliera G. Rummo, Benevento, BN
  - Ospedale Fatebenefratelli 'Sacro Cuore di Gesù', Benevento, BN
  - Presidio Ospedaliero 'Antonio Perrino', Brindisi, BR
  - ASST Spedali Civili - P.O. Spedali Civili, Brescia, BS
  - Ospedale Civile di Campobasso - A. Cardarelli, Campobasso, CB
  - Ospedale Vietri, Larino, CB
  - Ospedale Clinicizzato 'S. Annunziata' - Università degli Studi 'G. d'Annunzio', Chieti, CH
  - Ospedale Civile Renzetti, Lanciano, CH
  - Ospedale Civile 'Gaetano Bernabeo', Ortona, CH
  - Azienda Ospedaliera S. Croce e Carle, Cuneo, CN
  - ASST Lariana - Ospedale S. Anna, Como, CO
  - Humanitas Centro Catanese di Oncologia, Catania, CT
  - IRCCS Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.), Meldola, FC
  - Arcispedale S. Anna - A.O.U. di Ferrara, Cona, FE
  - IRCCS 'Casa Sollievo della Sofferenza', San Giovanni Rotondo, FG
  - A.O.U. Careggi, Florence, FI
  - AUSL di Frosinone - Ospedale Fabrizio Spaziani, Frosinone, FR
  - AUSL di Frosinone - Ospedale SS. Trinità, Sora, FR
  - IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy, Genoa, GE
  - E.O. Ospedali Galliera, Genova, GE
  - Azienda U.S.L. N. 9 - Ospedale Misericordia, Grosseto, GR
  - Azienda Sanitaria Regionale Molise - Ospedale F. Veneziale - Zona di Isernia, Isernia, IS
  - Ospedale Vito Fazzi, Lecce, LE
  - A.S.L. LT - Ospedale Santa Maria Goretti, Latina, LT
  - Ospedale Unico Versilia, Lido di Camaiore, LU
  - Ospedale San Luca, Lucca, LU
  - ASST Monza - Ospedale San Gerardo, Monza, MB
  - Ospedale di Macerata, Macerata, MC
  - ASST Melegnano e della Martesana - Ospedale Serbelloni, Gorgonzola, MI
  - ASST Ovest Milanese - Ospedale Nuovo di Legnano, Legnano, MI
  - ASST Fatebenefratelli Sacco - Ospedale Fatebenefratelli e Oftalmico, Milan, MI
  - Istituto Europeo di Oncologia (IRCCS), Milan, MI
  - Azienda Ospedaliera Carlo Poma, Mantova, MN
  - A.O.U. Policlinico Modena, Modena, MO
  - A.O.U. Policlinico 'Paolo Giaccone', Palermo, PA
  - Ospedale 'Guglielmo da Saliceto', Piacenza, PC
  - Istituto Oncologico Veneto - I.R.C.C.S., Padua, PD
  - Ospedale Civile 'San Massimo', Penne, PE
  - Ospedale Civile di Città di Castello - A.S.L. n. 1, Città di Castello, PG
  - Ospedale S. Maria della Misericordia, Perugia, PG
  - A.O.U. Pisana - Ospedale Santa Chiara, Pisa, PI
  - Ospedale Felice Lotti - Azienda USL 5 di Pisa, Pontedera, PI
  - Policlinico Umberto I, Roma, PM
  - Azienda Ospedaliera Universitaria di Parma, Parma, PR
  - Ospedale Santa Croce - A.O. Ospedali Riuniti Marche Nord, Fano, PS
  - Fondazione S. Maugeri IRCCS, Pavia, PV
  - Azienda Ospedaliera S. Carlo, Potenza, PZ
  - Ospedale per gli Infermi, Faenza, RA
  - Ospedale Umberto I, Lugo, RA
  - Azienda Ospedaliera Bianchi - Melacrino - Morelli, Reggio Calabria, RC
  - Ospedale San Sebastiano, Correggio, RE
  - Ospedale Civile di Guastalla, Guastalla, RE
  - IRCCS A.O. S.Maria Nuova, Reggio Emilia, RE
  - Istituto Regina Elena per lo studio e la cura dei tumori, Roma, RM
  - Ospedale S. Eugenio, Roma, RM
  - Azienda Ospedaliera San Camillo - Forlanini, Roma, RM
  - Ospedale Fatebenefratelli San Giovanni Calibita - Isola Tiberina, Roma, RM
  - A.O. S. Andrea - Università 'La Sapienza' - II Facoltà di Medicina e Chirurgia, Roma, RM
  - Azienda Ospedaliera n. 1 - Annunziata, Sassari, SS
  - Fondazione del Piemonte per l'Oncologia - IRCC di Candiolo, Candiolo, TO
  - Ospedale S. Anna - A.O.U. Città della Salute e della Scienza, Torino, TO
  - Ospedale S. Anna - Città della salute, Torino, TO
  - ASST della Valle Olona - Ospedale di Saronno, Saronno, VA
  - Ospedale Sacro Cuore Don Calabria, Negrar, VE
  - Ospedale Belcolle - AUSL di Viterbo, Viterbo, VT
  - A.O.U. Federico II, Napoli
  - Azienda Ospedaliera 'A. Cardarelli' (AORN), Napoli
  - Istituto Nazionale dei Tumori - Fondazione G.Pascale, Napoli

IPD SHARING:
Plan to Share IPD: No